CLINICAL TRIAL: NCT01085084
Title: A Phase IIa, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability and Clinical Effect of Laquinimod in Systemic Lupus Erythematosus Patients With Active Lupus Arthritis
Brief Title: A Study of Laquinimod in Participants With Systemic Lupus Erythematosus (SLE) Active Lupus Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LA-LAQ-202
Record Dates: First submitted 2010-03-09; First posted 2010-03-11 (Estimated); Results first posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-06

CONDITIONS: Lupus Arthritis
Keywords: Systemic Lupus Erythematosus (SLE); Lupus Arthritis; Laquinimod
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — laquinimod

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Participants will receive 2 capsules of placebo matched to laquinimod orally once daily for 12 weeks.
  Interventions: Drug: Placebo
- Laquinimod 0.5 mg (Experimental): Participants will receive 1 capsule of laquinimod 0.5 mg and 1 capsule of placebo matched to laquinimod orally once daily for 12 weeks.
  Interventions: Drug: Laquinimod; Drug: Placebo
- Laquinimod 1 mg (Experimental): Participants will receive 2 capsules of laquinimod 0.5 mg orally once daily for 12 weeks.
  Interventions: Drug: Laquinimod

INTERVENTIONS:
Drug: Laquinimod — Laquinimod will be administered per dose and schedule specified in the arm description.
  Arms: Laquinimod 0.5 mg; Laquinimod 1 mg
Drug: Placebo — Placebo matching to laquinimod will be administered per schedule specified in the arm description.
  Arms: Laquinimod 0.5 mg; Placebo

SUMMARY:
The study aims to evaluate the safety and clinical effect of daily oral treatment with laquinimod capsules (0.5 milligrams [mg] and 1 mg) in participants with active lupus arthritis. Laquinimod is a novel immunomodulating drug which is currently in advanced stages of development by Teva Pharmaceuticals Ltd. for Multiple Sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with SLE.
* Participants with active lupus arthritis as evident by at least 4 tender and 4 swollen joints at screening and baseline visits, and moderate or severe arthritis with active synovitis in at least 1 joint, with some loss of functional range of movement present at screening and baseline visits.

Exclusion Criteria:

* The participant's estimated glomerular filtration rate (eGFR) was less than or equal to 30 milliliters (mL)/minute/1.73 square meter (m^2), as calculated by the Modification of Diet in Renal Disease (MDRD) formula at the screening visit.
* Participants with severe, unstable and/or progressive central nervous system (CNS) lupus and/or associated with significant cognitive impairment (upon the investigators' judgement).
* Participants with a clinically significant or unstable medical or surgical condition that, in the investigator's opinion, would preclude safe and complete study participation.
* Women who are pregnant or nursing or who intend to be during the study period.
* Women of child-bearing potential who do not practice an acceptable method of birth control.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2010-10-04 (Actual); Primary Completion 2012-11-12 (Actual); Study Completion 2012-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, M.D., Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (22):
- United States (16):
  - Teva Investigational Site 1363, Birmingham, Alabama
  - Teva Investigational Site 1368, Los Angeles, California
  - Teva Investigational Site 1359, Los Angeles, California
  - Teva Investigational Site 1352, San Francisco, California
  - Teva Investigational Site 1365, San Leandro, California
  - Teva Investigational Site 1357, Stanford, California
  - Teva Investigational Site 1367, Chicago, Illinois
  - Teva Investigational Site 1370, Baltimore, Maryland
  - Teva Investigational Site 1362, Cumberland, Maryland
  - Teva Investigational Site 1360, Hagerstown, Maryland
  - Teva Investigational Site 1353, Manhasset, New York
  - Teva Investigational Site 1355, New York, New York
  - Teva Investigational Site 1369, The Bronx, New York
  - Teva Investigational Site 1356, Charlotte, North Carolina
  - Teva Investigational Site 1354, Columbus, Ohio
  - Teva Investigational Site 1366, Charleston, South Carolina
- Canada (6):
  - Teva Investigational Site 1139, Edmonton, Alberta
  - Teva Investigational Site 1141, Vancouver, British Columbia
  - Teva Investigational Site 1138, Winnipeg, Manitoba
  - Teva Investigational Site 1136, London, Ontario
  - Teva Investigational Site 1137, Toronto, Ontario
  - Teva Investigational Site 1142, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received 2 capsules of placebo matched to laquinimod orally once daily for 12 weeks.
- Laquinimod 0.5 mg: Participants received 1 capsule of laquinimod 0.5 milligrams (mg) and 1 capsule of placebo matched to laquinimod orally once daily for 12 weeks.
- Laquinimod 1 mg: Participants received 2 capsules of laquinimod 0.5 mg orally once daily for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | Laquinimod 0.5 mg | Laquinimod 1 mg
Started | 26 | 28 | 28
Received at Least 1 Dose of Study Drug | 26 | 28 | 28
Safety Analysis Set | 25 | 29 (1 participant was assigned to placebo but received laquinimod 0.5 mg by mistake.) | 28
Completed | 19 | 23 | 19
Not Completed | 7 | 5 | 9
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 1
Not completed — Adverse Event | 4 | 3 | 6
Not completed — Treatment Failure | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Intent-To-Treat (ITT) analysis set included all participants who were randomly assigned to a treatment, regardless of which treatment they actually received.
Groups:
- Laquinimod 0.5 mg: Participants received 1 capsule of laquinimod 0.5 mg and 1 capsule of placebo matched to laquinimod orally once daily for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Laquinimod 0.5 mg | Laquinimod 1 mg | Total
Number analyzed (Participants) | 26 | 28 | 28 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (13.5) | 46.6 (12.0) | 46.8 (13.4) | 47.1 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 25 | 26 | 75
  Male | 2 | 3 | 2 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 2 | 0 | 2
  Black or African American | 4 | 3 | 9 | 16
  White | 16 | 14 | 10 | 40
  Hispanic | 6 | 8 | 8 | 22
  Native Hawaiian or Pacific Islander | 0 | 1 | 0 | 1
  Other | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both SAEs and non-serious AEs. A summary of other non-serious AEs and all SAEs, regardless of causality is located in the 'Reported AE section'.
Time Frame: Baseline up to Week 16
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug. In this set, treatment was assigned based upon the treatment actually received regardless of the assigned treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Laquinimod 0.5 mg | Laquinimod 1 mg
Number analyzed (Participants) | 25 | 29 | 28
Participants | 21 | 29 | 25

2. Primary Outcome: Percent Change From Baseline in Swollen Joint Count at Week 12
Description: The number of swollen joints was used to assess lupus arthritis activity. Joint swelling was defined as soft tissue swelling that was detectable along the joint margins. 66 joints were examined for swelling. These joints include the temporomandibular (n = 2), sternoclavicular (n =2), acromioclavicular (n = 2), shoulder (n = 2), elbow (n = 2), wrist (n = 2), metacarpophalageal (n= 10), interphalangeal of thumb (n = 2), distal interphalangeal (n = 8), proximal interphalangeal (n =8), knee (n = 2), ankle mortise (n = 2), ankle tarsus (n = 2), metatarsophalangeal (n = 10), interphalangeal of great toe (n = 2), and proximal/distal interphalangeal of the toes (n = 8).
Time Frame: Baseline, Week 12
Population: Modified intent-to-treat (mITT) analysis set included all participants who were randomly assigned to a treatment, regardless of which treatment they actually received, excluding observations after treatment failure. Here 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Laquinimod 0.5 mg | Laquinimod 1 mg
Number analyzed (Participants) | 26 | 27 | 26
percent change | -36.9 (78.1) | -36.7 (47.0) | -40.5 (55.6)

3. Primary Outcome: Percent Change From Baseline in Tender Joint Count at Week 12
Description: The number of tender joints was used to assess lupus arthritis activity. Joint tenderness was defined as the presence or absence of tenderness and/or pain in a joint at rest with pressure or on passive movement of the joint and joint manipulation. 68 joints were examined for tenderness. These joints include the temporomandibular (n = 2), sternoclavicular (n =2), acromioclavicular (n = 2), shoulder (n = 2), elbow (n = 2), wrist (n = 2), metacarpophalageal (n= 10), interphalangeal of thumb (n = 2), distal interphalangeal (n = 8), proximal interphalangeal (n =8), hip (n = 2), knee (n = 2), ankle mortise (n = 2), ankle tarsus (n = 2), metatarsophalangeal (n = 10), interphalangeal of great toe (n = 2), and proximal/distal interphalangeal of the toes (n = 8).
Time Frame: Baseline, Week 12
Population: The mITT analysis set included all participants who were randomly assigned to a treatment, regardless of which treatment they actually received, excluding observations after treatment failure. Here 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Laquinimod 0.5 mg | Laquinimod 1 mg
Number analyzed (Participants) | 26 | 27 | 26
percent change | -8.5 (81.3) | -31.4 (53.1) | -42.0 (37.8)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 16
Description: Safety analysis set included all randomized participants who received at least 1 dose of study drug. In this set, treatment was assigned based upon the treatment actually received regardless of the assigned treatment.
Arm/Group | Placebo | Laquinimod 0.5 mg | Laquinimod 1 mg
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/29 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/25 | 4/29 | 2/28
Other Adverse Events (participants affected / at risk) | 17/25 | 24/29 | 18/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=25) | Laquinimod 0.5 mg (N=29) | Laquinimod 1 mg (N=28)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia Mycoplasmal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=25) | Laquinimod 0.5 mg (N=29) | Laquinimod 1 mg (N=28)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (4)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2)
Abdominal Tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 4 (4) | 4 (5)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3) | 5 (7) | 6 (6)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (4) | 2 (2)
Fatigue (General disorders) | 2 (2) | 1 (1) | 3 (4)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 2 (2)
Seasonal Allergy (Immune system disorders) | 0 (0) | 0 (0) | 2 (2)
Escherichia Urinary Tract Infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Tooth Infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 4 (5) | 2 (3)
Urinary Tract Infection (Infections and infestations) | 4 (7) | 1 (1) | 2 (2)
Muscle Strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (4)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Systemic Lupus Erythematosus (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 4 (5) | 3 (5)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.